CLINICAL TRIAL: NCT05557604
Title: Sbrt±sTad for Unfavorable iNtermediate rIsk/High Risk Prostate caNcer (STUNNIN): A Randomized Phase II Study
Brief Title: Sbrt±sTad for Unfavorable iNtermediate rIsk/High Risk Prostate caNcer
Acronym: STUNNIN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Regina Elena Cancer Institute (Other)
Responsible Party: Principal Investigator, Giuseppe Sanguineti, Professore, Regina Elena Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RS1399/20(2384) PU
Record Dates: First submitted 2022-09-23; First posted 2022-09-28 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Prostate Cancer
Keywords: neoplasm, prostate cancer,
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Triptorelin Pamoate; Leuprolide

STUDY DESIGN:
Intervention Model Description: prospective, open, randomized phase 2 trial
Who Masked: Investigator
Masking Description: Subjects who meet all study eligibility criteria will be randomly assigned in a 1:1 ratio.
  Randomization is centralized at the promoter and takes place according to a specific procedure (in attachment).
  The randomization schedule will be generated by an independent group of the promoter.
  Patient study number and result of randomization will be given immediately by email.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- arm 1 (No Intervention): SBRT alone 38 GY in 4 fractions
- arm 2 (Experimental): SBRT along with short course (6 months) androgen deprivation (STAD)
  Interventions: Drug: Decapeptyl

INTERVENTIONS:
Drug: Decapeptyl — STAD androgen deprivation
  Other Names: Enantone
  Arms: arm 2

SUMMARY:
This is a prospective, open, randomized phase II trial.

DETAILED DESCRIPTION:
Patients will be randomized between SBRT alone (38 Gy in 4 fractions) or SBRT (same schedule) along with short course (6 months) androgen deprivation (STAD). All patients will be treated by intensity modulated radiotherapy. Regarding the combined modality approach, SBRT has to start within 3 months from the first injection of LHRH analogue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate adenocarcinoma
* IR or HR in the NCCN definition
* N0M0 at staging with choline or (preferably) PSMA PET-CT;
* ECOG performance status between 0 and 2;

Exclusion Criteria:

* Previous local treatment of the prostate with surgery (radical prostatectomy or cryotherapy)
* Previous radiotherapy to the pelvis
* Previous chemotherapy for malignancy in past 5 years
* Impossibility to implant fiducials for tracking purposes
* Impossibility to undergo MRI of the prostate
* Contraindication to short term AD
* Prostate volume >90cc

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2021-02-02 (Actual); Primary Completion 2024-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
3-yr bNED survival | 3 years
  The primary objective of the study is 3-yr bNED survival. If bNED survival is not significantly different between the two experimental arms, the one without AD will be chosen in a future comparison with the standard of care.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Ifo Regina elena, Rome, Lazio
  - ifo Regina Elena, Rome, RM
  - Regina Elena National Cancer Institute, Rome